CLINICAL TRIAL: NCT00765609
Title: To Evaluate the Paediatric Analgesia Slide, a New Device Developed to Assist Parents in Administering Paracetamol to Children at Home
Brief Title: To Evaluate the Paediatric Analgesia Slide
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: County Durham and Darlington NHS Foundation Trust (Other Government)
Responsible Party: Dr Richard Hixson, County Durham and Darlington NHS Foundation Trust
Other Study IDs: 08/H0904/93
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-09

CONDITIONS: Pain
Keywords: Paediatric; Analgesic; Prescribing; Parents
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Using the information distributed with over-the-counter medication (The Patient Information Leaflet or PIL)
- 2: Paediatric Analgesia Slide (the new device)

SUMMARY:
The Paediatric Analgesia Slide is a device developed for parents. Its development follows research into the Paediatric Analgesia Wheel, a device intended for use by hospital doctors. Previous research has shown the benefit of using aids such as the Paediatric Analgesia Wheel when simulating prescribing to children in hospital.

At present, it is unknown whether this concept can be extended to use by parents when administering paracetamol to their children at home.

DETAILED DESCRIPTION:
Prescribing and administering drugs to children is difficult for both healthcare professionals and parents. The process is often performed poorly with under-dosing and over-dosing a major problem with sometimes fatal consequences.

The British National Formulary for Children (BNFC), introduced in 2005, has given hospital and community prescribers with a valuable reference text.

However, the comprehensive prescribing information presented in the BNFC and in the drug Summary of Product Characteristics is simplified in the Patient Information Leaflet (PIL) for interpretation by parents. When the PIL is analysed, it becomes apparent that the age-range regimens presented may result in under and over-dosing with large differences in the daily dose received by children depending on their age and weight.

The Paediatric Analgesia Slide is a simple device presenting pre-calculated volume (and therefore dose) information for parents. It allows for age/weight specific doses to be given thus minimising the risk of under and over-dosing. It also addresses the deficiency of the prescribing information in the PIL related to over and under-weight children.

ELIGIBILITY:
Inclusion Criteria:

* Any parent accompanying their child who is aged between 1 and 13 years old who is attending a hospital in County Durham and Darlington Acute Hospitals NHS Trust

Exclusion Criteria:

* Those who have professional knowledge of prescribing or dispensing medicine (e.g. as a doctor, nurse or pharmacist);
* Those who already have been given advice on the correct dose of paracetamol for their child as part of the current hospital episode;
* Those who's child is under 1 year or over 13 years old and;
* Those who have participated in this research before.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: parents administering analgesic medication to their children
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-02 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of prescription accuracy using the information distributed with over-the-counter medication with the new device | at data analysis

SECONDARY OUTCOMES:
Ability of parents to interpret the prescribing information related to minimum dosage interval and maximum dosage frequency | at data analysis
To assess whether parents can accurately draw up the volume that they have stated in the primary objective | at data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Hixson, BM BS, FRCA, Principal Investigator — County Durham and Darlington Acute Hospitals NHS Trust
Locations (1):
- County Durham and Darlington Acute Hospitals NHS Trust, Darlington, England, United Kingdom